CLINICAL TRIAL: NCT06712212
Title: Non-mesh Repair of Inguinal Hernia: Desarda Versus Darn
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Akram Hamad, Resident General Surgery, Assiut University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Inguinal hernia repair
Record Dates: First submitted 2024-09-27; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Inguinal Hernia Repair; Inguinal Hernia
Keywords: Hernia; Desarda repair; Darn repair; Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal; Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Inguinal hernia (Active Comparator)
  Interventions: Procedure: Inguinal Hernias repair: Desarda; Procedure: Inguinal hernia repair: Darn

INTERVENTIONS:
Procedure: Inguinal Hernias repair: Desarda — A splitting incision is made in this sutured medial leaf, partially separating a strip 1.5-2 cm wide. This splitting incision is extended medially up to the pubic symphysis and 1-2 cm beyond the abdominal ring laterally. The medial insertion and lateral continuation of this strip is kept intact. The upper free border of the strip is now sutured to the internal oblique with number 1 Monofilament Polydioxanone Violet continuous sutures all along its length. This will result in the strip of the EOA being placed behind the cord to form a new posterior wall of the inguinal canal. The spermatic cord is placed in the inguinal canal and the lateral leaf of the EOA is sutured to the newly formed medial leaf of the EOA in front of the cord. As before, number 1 Monofilament Polydioxanone Violet continuous sutures were used. Undermining of the newly formed medial leaf on both its surfaces and excision of the bulky cremasteric muscle facilitate its approximation to the lateral leaf
  Other Names: Desarda repair of inguinal hernia
Procedure: Inguinal hernia repair: Darn — Skin and fascia are incised using a regular, oblique inguinal incision to expose the external oblique aponeurosis (EOA) the inguinal canal is opened into by dividing the external oblique aponeurosis through the external ring. After dealing with the hernia sac, a 0-size monofilament suture was used to reconstruct the inguinal bed with a tension-free darn starting with a good strong bite of the tough tendinous structures near the pubic tubercle and emerging out through the lateral edge of the internal oblique/rectus sheath from one side and through the inguinal ligament on the other side. The loosely interwoven bites continued laterally and the back-forming two rows of continuous stitches were placed in a staggered manner to spread the tension between the fibres of the inguinal ligament. Afterwards, the external oblique and other superficial layers with the skin are classically closed
  Other Names: Darn repair of inguinal hernia

SUMMARY:
To compare the results of Desarda and Darn techniques in inguinal hernia repair in Assiut University Hospital.

DETAILED DESCRIPTION:
Inguinal hernia is one of the most common types of abdominal hernias with a prevalence of 75% of all abdominal hernias. Inguinal hernia repair is one of the most encountered surgeries all over the world. The use of mesh for inguinal hernia repair is the most commonly applied technique. However, being a foreign body, mesh repair has its own disadvantages. These include Postoperative hematoma and seroma, foreign body reaction, infection, mesh rejection, mesh migration, and fistula formation. Moreover, the use of mesh in potentially contaminated operating field is not advisable. Infectious complication and their consequences have restricted the use of mesh in emergency settings. In addition, mesh repair is not available in every part of the world since it increases the cost of the operation. Therefore, the non-mesh repair of inguinal hernia has been recently revisited. Different techniques for non-mesh inguinal hernia repair are available including Bassini, Shouldice, Desarda and Darn. In 2001,Indian Surgeon Dr. Desarda, introduced a novel technique of a tissue- based hernia repair without mesh with almost zero recurrence rates in which an undetached strip of the external oblique aponeurosis is sutured to the inguinal ligament below and the muscle arch above, behind the cord, to form a new posterior wall. External oblique muscle gives additional strength to the weakened muscle arch to keep this strip physiologically dynamic. In 1948, Moloney described a suture inguinal herniorrhaphy in which two layers of continuous monofilament non-absorbable suture lines with no tension were inserted. The first suture line is between the lower edge of the internal oblique muscle/aponeurosis and the inguinal ligament. The second superficial layer is between the rectus sheath and the inguinal ligament. All sutures should be placed without tension but with no slack .

Literature are deficient in comparing Desarda technique and Darn technique in the repair of inguinal hernia.

ELIGIBILITY:
Inclusion Criteria:

* inguinal hernia
* Age more than 18
* Male patients

Exclusion Criteria:

• simultaneous performance of other surgical procedures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Short term recurrence of hernia | From the day post operative to 6 months after the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided